CLINICAL TRIAL: NCT04261959
Title: Longitudinal Analysis of an Innovative Non-Pharmacological Intervention for Chronic Pain in a Marginalized Population: A Prospective Pilot Study of myoActivation
Brief Title: myoActivation® for Chronic Pain in a Marginalized Population
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other); BC Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Barbara Eddy, Associate Member in the UBC Department of Medicine, Division of Palliative Care, University of British Columbia
Other Study IDs: H19-02567
Record Dates: First submitted 2020-02-03; First posted 2020-02-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2022-11

CONDITIONS: Pain, Chronic; Widespread Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- myoActivation and other pain services: Participants who receive one or more sessions of myoActivation. They may receive 1:1 counselling and physiotherapy also.
  Interventions: Other: myoActivation

INTERVENTIONS:
Other: myoActivation — myoActivation is a novel, structured assessment and non-pharmacological therapeutic approach to both diagnosis and treatment of chronic myofascial pain. A detailed history of the timeline of lifetime trauma combined with a quick, structured and reproducible set of posture and movement tests help to easily identify myofascial components of chronic pain. The therapeutic component is delivered utilizing a needling technique, or myofascial release, focused to active myofascial trigger points, fascia in tension and tethered scars.

SUMMARY:
Marginalized populations are at increased risk of chronic pain, trauma and use of street drugs to manage this suffering, with the associated risk of overdoses. Non-pharmacological options to manage chronic pain are difficult for this population to access. myoActivation® is an innovative structured assessment and therapeutic approach. This study will be conducted in the Vancouver Community Pain Service and will will examine the impact of this treatment on pain outcomes, function and quality of life.

DETAILED DESCRIPTION:
Purpose: This study will evaluate the inclusion of myoActivation in primary care for marginalized persons with concurrent opioid use disorder (OUD), chronic pain and trauma history. The research aims to investigate whether myoActivation improves pain intensity, quality of life, physical function, and reduces the need for prescribed analgesics (including opioids) and reported illicit drug use.

Hypothesis: The investigators hypothesize that patients with chronic pain who are treated with myoActivation will experience a reduction in pain and improvement in function and quality of life as shown by a 30% reduction on the PEG score (Pain intensity, interference with Enjoyment of life, interference with General activity) at 4, 12 and 24 weeks.

Justification: Chronic pain is typically treated by prescription of analgesic medications, including opioids. However, many patients who have overdoses are using opioids and other substances (including street drugs, alcohol, and marijuana) to manage chronic pain. There are an inadequate number of effective non-pharmacological options to manage chronic pain and wait lists for local Vancouver chronic pain clinics are as long as a year. Other treatment modalities offered by the Vancouver Community pain service include physiotherapy and counselling.

Objectives: The investigators aim to demonstrate an improvement in pain intensity, quality of life, and physical function as the primary outcomes. Secondary objectives include reduced need for analgesic medications (including opioids) and illicit drug use.

Research Design: This study is a prospective, mixed method design, including 1:1 semi-structured patient interviews. It is an observational study: patients will NOT be allocated to treatment on the basis of randomization or their enrollment in the study, i.e. participants will receive routine clinical care, based on the services offered by the clinical team at the pain clinic, and this will not change with their participation in the study.

The study will involve recruitment of 40 patients who attend the pain service on Tuesdays, when myoActivation and physiotherapy are offered, and who consent to being contacted for follow up data collection and interviews. At the time of recruitment, the subset of patients who have concurrent opioid use disorder, other addictions and / or trauma will not be known.

Data collection includes:

* a baseline score of the patients' pain experience using the validated questionnaires PEG, Pain Catastrophizing Scale (PCS) and Pain Self-Efficacy Questionnaire (PSEQ).
* information on baseline mental health conditions - OUD, Trauma, Anxiety, Depression, Axis 1
* PEG, PCS, PSEQ scores as well as the patient reported use of street drugs and pain medications will be collected at 4, 12, 24 weeks using a study designed questionnaire
* a semi-structured 1:1 patient interview at 12-24 weeks will assess opioid/drug use, as well as questions related to changes to housing, finances and overall health; this will be conducted with 10 randomly selected participants who have received myoActivation.

Statistical Analysis: To allow for correlation of repeated data points on the same patient as well as the anticipated variability in the number of data points for each patient, a linear mixed-effects model will be used to analyze the quantitative data, including PEG score and self-reported opioid use. A PEG score decrease of 30% will be taken to indicate an improved pain experience. The PCS and PSEQ scores will be used to interpret the severity and change of an individual's pain score.

The patient interview responses will be collated for common themes and used to augment the quantitative data outcomes. Interviews will be recorded and transcribed. Thematic analysis will be used to identify key words and phrases, list noted benefits of the service, potential problems raised and any preferences expressed by participants with respect to the way the treatment is administered.

ELIGIBILITY:
Inclusion Criteria:

Any English-speaking patient with myofascial related chronic pain lasting >3 months, referred to the Vancouver Community (VC) chronic pain service by primary care.

Exclusion Criteria:

Any patient who has received any of the following pain interventions or treatment in the 3 months preceding recruitment/intake to the pain service:

* Intramuscular Stimulation (IMS);
* Trigger Point Injection (TPI) with or without injectate;
* External physiotherapy (i.e. outside the service offered at VC pain clinic);
* Massage;
* Joint injection;
* Chiropractic;
* Acupuncture;
* Group counselling at VC Pain Service (or has an existing appointment to attend Group counselling).

(note, exclusion list does not include pain medications or opioid replacement therapy; also note, patients who subsequently access the VC Pain Service Group counselling will continue to be included in the study)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Structurally vulnerable persons (i.e. within marginalized populations) with chronic pain, and typically also mental health issues, substance use disorders, physical and emotional trauma.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
PEG score wk 4 | 4 weeks
  PEG is a validated self-report measure of (1) Pain intensity, (2) interference with Enjoyment of life, (3) interference with General activity. Each of the 3 dimensions is scored on a 0-10 scale. Total score is the average (mean) of the 3 values, minimum 0, maximum 10, lower score indicates a better outcome.
PEG score wk 12 | 12 weeks
  PEG is a validated self-report measure of (1) Pain intensity, (2) interference with Enjoyment of life, (3) interference with General activity. Each of the 3 dimensions is scored on a 0-10 scale. Total score is the average (mean) of the 3 values, minimum 0, maximum 10, lower score indicates a better outcome.
PEG score wk 24 | 24 weeks
  PEG is a validated self-report measure of (1) Pain intensity, (2) interference with Enjoyment of life, (3) interference with General activity. Each of the 3 dimensions is scored on a 0-10 scale. Total score is the average (mean) of the 3 values, minimum 0, maximum 10, lower score indicates a better outcome.

SECONDARY OUTCOMES:
PCS score wk 4 | 4 weeks
  Pain Catastrophizing Scale (PCS) is a validated self-report scale that measures a person's cognitive-affective response to pain including the person's sense of helplessness, rumination and magnification of pain. Each of 13 dimensions are scored 0-4. The total score is the sum of these dimensions, minimum 0, maximum 52, lower score indicates a better outcome.
PCS score wk 12 | 12 weeks
  Pain Catastrophizing Scale (PCS) is a validated self-report scale that measures a person's cognitive-affective response to pain including the person's sense of helplessness, rumination and magnification of pain. Each of 13 dimensions are scored 0-4. The total score is the sum of these dimensions, minimum 0, maximum 52, lower score indicates a better outcome.
PCS score wk 24 | 24 weeks
  Pain Catastrophizing Scale (PCS) is a validated self-report scale that measures a person's cognitive-affective response to pain including the person's sense of helplessness, rumination and magnification of pain. Each of 13 dimensions are scored 0-4. The total score is the sum of these dimensions, minimum 0, maximum 52, lower score indicates a better outcome.
PSEQ score wk 4 | 4 weeks
  Pain Self-Efficacy Questionnaire (PSEQ) is a validated self-report scale, designed to assess the confidence people with ongoing pain have in performing activities while in pain. Each of 4 dimensions is scored 0-6. The total score is the sum of these dimensions, minimum 0, maximum 24, lower score indicates a worse outcome.
PSEQ score wk 12 | 12 weeks
  Pain Self-Efficacy Questionnaire (PSEQ) is a validated self-report scale, designed to assess the confidence people with ongoing pain have in performing activities while in pain. Each of 4 dimensions is scored 0-6. The total score is the sum of these dimensions, minimum 0, maximum 24, lower score indicates a worse outcome.
PSEQ score wk 24 | 24 weeks
  Pain Self-Efficacy Questionnaire (PSEQ) is a validated self-report scale, designed to assess the confidence people with ongoing pain have in performing activities while in pain. Each of 4 dimensions is scored 0-6. The total score is the sum of these dimensions, minimum 0, maximum 24, lower score indicates a worse outcome.
Drug use wk 4 | 4 weeks
  Patient reported use of street drugs and pain medications; whether participant is on opioid replacement therapy currently, or in the past.
Drug use wk 12 | 12 weeks
  Patient reported use of street drugs and pain medications; whether participant is on opioid replacement therapy currently, or in the past.
Drug use wk 24 | 24 weeks
  Patient reported use of street drugs and pain medications; whether participant is on opioid replacement therapy currently, or in the past.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Eddy, Principal Investigator — Vancouver Coastal Health
Locations (1):
- Vancouver Community Pain Service, 524 East Pender Street, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen L, Eddy BL, West N, Bone JN, Currie LM, Lauder G. The Impact of a Novel Methodological Process for Needling Scars, Fascia, and Muscles in the Management of Myofascial Dysfunction and Chronic Pain in a Population Living With Social and Health Inequities: Quantitative Findings From a Longitudinal Observational Pilot Study. Pain Res Manag. 2025 Sep 28;2025:8567447. doi: 10.1155/prm/8567447. eCollection 2025. PMID 41058955